CLINICAL TRIAL: NCT04138576
Title: Evaluation of the Efficacy and Tolerability of Venoactive Drugs in Combination Therapy and Their Effect on the Overall Treatment Outcomes in Patients With Chronic Venous Diseases of CEAP Class C4a and C4b in Real Clinical Practice.
Brief Title: Efficacy and Tolerability of Venoactive Drugs in Patients With Chronic Venous Diseases C4a&b in Real Clinical Practice.
Acronym: VAP-PRO-C4
Status: Completed | Type: Observational
Sponsor: Servier Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4-05682-059-RUS
Record Dates: First submitted 2019-10-16; First posted 2019-10-24 (Actual); Results first posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-10

CONDITIONS: Chronic Venous Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is aimed at evaluating the efficacy and tolerability of systemic pharmacotherapy as a part of combination treatment, and its influence on the overall treatment outcomes in patients with skin changes (CEAP class C4a and C4b).

DETAILED DESCRIPTION:
Primary goal:

To study the efficacy of systemic pharmacotherapy as part of combination therapy and its impact on the:

* thickness of the skin-fat fold (ultrasound examination);
* change in the venous clinical severity score (VCSS);
* change in the CEAP clinical class of CVD;
* evolution of CVD symptoms characteristic for CEAP class C4 (sensations of skin tightening, burning, itching, pain, and exudation) using the Visual Analogue Scale (VAS).

Secondary goals:

1. To study the efficacy of systemic pharmacotherapy as part of combination therapy and its impact on the:

   * area of affected skin determined by curvimetry technique (only in selected centers that use this technique routinely) before and after the treatment in patients with skin changes of CEAP class C4a or C4b in real clinical practice;
   * skin density determined by durometry technique (only in selected centers that use this technique routinely).
2. To evaluate the changes in the quality of life using the CIVIQ-14 questionnaire (global index score [GIS]) .
3. To study the tolerability of systemic pharmacotherapy as part of combination therapy in patients with skin changes of CEAP class C4a or C4b.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or above
* Written informed consent
* Patient did not receive treatment with venoactive drugs within the past 4 -weeks prior to the inclusion in the study
* Diagnosis of chronic venous disease of CEAP class C4
* No surgical intervention for CVD is planned by a doctor

Exclusion Criteria:

* Chronic venous disease of СЕАР class C0-С3 or class С4-С6
* History of alcohol or drug abuse or use of narcotic drugs
* Peripheral artery disease
* Lymphatic edema of the lower extremities
* Secondary varicose veins, angiodysplasia, or neoplasia
* Arterial disease (ankle-brachial index <0.9)
* Infection within the past 6 weeks
* Any of the following concomitant diseases, which can affect the results:
* Connective tissue disease (including rheumatoid arthritis), arthritis
* Heart failure
* Chronic kidney disease
* Decompensated diabetes mellitus
* Skin diseases of non-venous origin
* Intermittent claudication (peripheral artery disease)
* Diseases of the bones or joints of the lower extremities
* Malignancy

Treatment with drugs potentially causing leg edema (calcium channel blockers, hormonal drugs, NSAIDs, etc.) History of deep vein thrombosis (within the past year) History of superficial thrombophlebitis (within the past 3 months) History of surgical intervention (within the past 3 months) Patient cannot walk (regardless of the cause) Predictable poor adherence to treatment Participation of a patient in the intervention study within the previous 3 months For women: pregnancy or breastfeeding, the desire to become pregnant within at least 2 months after the study Patients with a contraindication to diosmin-containing agents, including Detralex Patient uses the topical treatments contraindicated in case of skin integrity violation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic venous diseases of CEAP class C4a and C4b
Sampling Method: Non-Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Linnik, Study Chair — Medical manager
Locations (1):
- National Medical and Surgical Center. N.I. Pirogov, Moscow, Russia

REFERENCES:
- [Derived] Bogachev V, Boldin B, Turkin P, Samenkov A, Dzhenina O. Micronized purified flavonoid fraction-based conservative treatment of chronic venous disease in a real-world setting. Future Cardiol. 2022 Sep;18(10):777-785. doi: 10.2217/fca-2022-0026. Epub 2022 Aug 25. PMID 36004765

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice: The study enrolled adults (≥18 years old) with CVD of CEAP class C4 (a or b) severity whose physicians recommended the initiation of MPFF (1000 mg/day) in addition to conservative treatment according to routine clinical practice, and for whom surgical intervention for their CVD was not currently planned
Period: Overall Study
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
Started | 381
Completed | 365
Not Completed | 16
Not completed — Due to epidemiological situation (COVID-19) patients were dropped out from the study. | 16

BASELINE CHARACTERISTICS:
Groups:
- Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice: According to the international CEAP classification, chronic venous diseases of clinical class C4 are characterized by various changes of skin and subcutaneous tissue of the affected limbs. They include skin hemosiderosis, Milian's white atrophy, indurative cellulitis, lipodermatosclerosis, and varicose eczema.
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
Number analyzed (Participants) | 365
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 269
  >=65 years | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.24 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239
  Male | 126
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 365
Patients with chronic venous diseases of CEAP classes C4a and C4b in real clinical practice [Count of Participants; unit: Participants] | 365

OUTCOME MEASURES:

1. Primary Outcome: The Mean Subcutaneous Adipose Tissue Thickness Changes (mm) Between the Visit 3 and Baseline by Ultrasound Examination.
Description: Ultrasound examination was used to get:
  1. Thickness of the thickness of the skin-fat fold at the affected skin area;
  2. Presence of reflux or occlusion (with an indication of the terrotiry).
     * Measurements should be taken in the afternoon at about the same time, at visits V0 and V3.
     * The data are recorded only for the limb with the most severe changes.
     * Measurements are taken at the site of skin changes. Unit of Measure - mm
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
Number analyzed (Participants) | 365
mm | 2.5 (4.5)

2. Secondary Outcome: The Mean Changes VCSS for Pain (Four-point Scale (From 0 to 3)) Between the Visit 3 and Baseline by Ultrasound Examination. Change in the VCSS Scale
Description: Was used four-point scale the Venous Clinical Severity Score(VCSS ). It uses a number of clinical signs, which are assigned a point equivalent depending on their severity (pain, varicose veins, edema, hyperpigmentation, inflammation, induration, the number of ulcers, the presence of active ulcers, the use of compression therapy). The sum of points reflects the severity of the pathology: the more points, the more severe the course of chronic venous disease. Changing the amount of points over time allows you to assess the degree of disease progression or the effectiveness of treatment measures.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: point on scale
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
Number analyzed (Participants) | 365
point on scale | 0.74 (0.68)

3. Secondary Outcome: The Mean Changes VCSS for Hyperpigmentation (Four-point Scale (From 0 to 3)) Between the Visit 3 and Baseline by Ultrasound Examination. Change in the VCSS Scale
Description: as for outcome 2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: point on scale
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
Number analyzed (Participants) | 365
point on scale | 0.49 (0.74)

4. Secondary Outcome: The Mean Changes VCSS for Inflammation (Four-point Scale (From 0 to 3)) Between the Visit 3 and Baseline by Ultrasound Examination. Change in the VCSS Scale
Description: as for outcome 2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: point on scale
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
Number analyzed (Participants) | 365
point on scale | 0.45 (0.74)

5. Secondary Outcome: Outcome Measure Title: The Mean Changes VCSS for Subcutaneous Tissue Induration (Four-point Scale (From 0 to 3)) Between the Visit 3 and Baseline by Ultrasound Examination. Change in the VCSS Scale
Description: as for outcome 2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: point on scale
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
Number analyzed (Participants) | 365
point on scale | 0.36 (0.71)

6. Secondary Outcome: The Mean CVD Symptoms Characteristic Changes Between the Visit 3 and Baseline Evaluated by Means of Visual Analogue Scale (VAS). -Skin Tightening
Description: Visual Analogue Scale (VAS) The Visual Analogue Scale (VAS) is designed to measure symptom's intensity. It is a continuous scale in the form of a horizontal or vertical line 10 cm (100 mm) long with two extreme points located on it: "no symptom " and "the strongest symptom you can imagine."
  Visual analogue scale technique:
  The patient is asked to place a line perpendicularly crossing the visual analogue scale at the point that corresponds to his symptom intensity. The ruler measures the distance (mm) between "no symptom" and "the worst symptom imaginable," providing a score range of 0 to 100. A higher score indicates more pain intensity.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: point on scale
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
Number analyzed (Participants) | 365
point on scale | 2.63 (2.41)

7. Secondary Outcome: The Mean CVD Symptoms Characteristic Changes Between the Visit 3 and Baseline Evaluated by Means of Visual Analogue Scale (VAS). - Intensity of Burning Sensation
Description: as for outcome 6
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: point on scale
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
Number analyzed (Participants) | 365
point on scale | 2.40 (2.40)

8. Secondary Outcome: The Mean CVD Symptoms Characteristic Changes Between the Visit 3 and Baseline Evaluated by Means of Visual Analogue Scale (VAS). - Skin Itching
Description: as for outcome 6
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: point on a scale
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
Number analyzed (Participants) | 365
point on a scale | 2.66 (2.42)

9. Secondary Outcome: The Mean CVD Symptoms Characteristic Changes Between the Visit 3 and Baseline Evaluated by Means of Visual Analogue Scale (VAS). - Pain
Description: as for outcome 6
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: point on a scale
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
Number analyzed (Participants) | 365
point on a scale | 2.90 (2.33)

10. Secondary Outcome: The Mean CVD Symptoms Characteristic Changes Between the Visit 3 and Baseline Evaluated by Means of Visual Analogue Scale (VAS). - Exudation
Description: as for outcome 6
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: point on a scale
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
Number analyzed (Participants) | 365
point on a scale | 0.48 (1.45)

11. Secondary Outcome: The Mean Changes of Global Index CIVIQ-14 Score (GIS) Between the Visit 3 and Baseline Evaluated
Description: CIVIQ-14 - Chronic Venous Insufficiency Questionnaire (CIVIQ-14) is a specific questionnaire for venous disease. It was used to evaluate the changes in the quality of life (global index score - GIS) There are 14 questions in the CIVIQ-14, each with 5 possible answers (1 to 5), the minimum possible score being 14 and the maximum 70. In order to calculate the GIS, the difference between the final score and the minimum possible score is to be divided by the difference between the theoretical maximum and minimum scores (70-14=56), multiplied by 100.
  GIS = ([Final score - minimal possible score] / [Theoretical maximal - minimal score]) x 100 GIS = ([Final score - minimal possible score] / 56) x 100 GIS = ([Final score - 14] / 56) x 100 The least GIS corresponds with the best quality of life, the largest GIS corresponds with the worst.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Global Index CIVIQ-14 Score
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
Number analyzed (Participants) | 365
Global Index CIVIQ-14 Score | 22.4 (16.5)

12. Secondary Outcome: The Mean Lesion Area Changes Between the Visit 3 and Baseline Evaluated by Curvimetry Technique
Description: This technique was used in only in Selected Centers That Use This Technique Routinely:
  technique is measured length of the border of modified skin, using a measuring device called a curvimetr.
  The quality of treatment is assessed by comparing data on Visit 0 and Visit 3 Measurements are carried out 2 times on Visit 0 and Visit 3 (before and after the treatment) in patients with skin changes of CEAP class C4a or C4b A decrease in the figure value (in centimeters) on Visit 3 vs baseline means a good treatment result.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: centimeter
Groups:
- Patients With CVD of CEAP Classes C4a and C4b Included in Curvimetry Technique Group: (only in Selected Centers That Use This Technique Routinely).
Arm/Group | Patients With CVD of CEAP Classes C4a and C4b Included in Curvimetry Technique Group
Number analyzed (Participants) | 60
centimeter | 6.9 (13.4)

13. Secondary Outcome: The Mean Changes of the Skin Density Determined by Durometry Technique Between the Visit 3 and Baseline Evaluated.
Description: Shore Hardness scales is a scale for measuring the hardness of different materials.Total score has a range from 0 (the softest material) to 100 scores (the hardest material). Measurement was performed by Shore durometer (a device for measuring the hardness of a material). The method and scale were proposed by Albert F. Shore.
  This technique was used in only in Selected Centers That Use This Technique Routinely:
  technique: repeated measures to compare the scores before and after the treatment.
  Shore hardness is one of the methods for measuring the hardness of materials. In medicine, it is used to determine the density of the skin. In this study, the method was used to determine the density of the skin in the area of skin lesions in patients with CVD stage C4 (CEAP)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Patients With CVD of CEAP Classes C4a and C4b Included in Durometry Technique Group: durometry technique is ..... Was applied only in selected Centers that use this technique routinely.
Arm/Group | Patients With CVD of CEAP Classes C4a and C4b Included in Durometry Technique Group
Number analyzed (Participants) | 55
scores on a scale | 3.9 (9.3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Patients With Chronic Venous Diseases of CEAP Classes C4a and C4b in Real Clinical Practice
All-Cause Mortality (participants affected / at risk) | 0/381
Serious Adverse Events (participants affected / at risk) | 0/381
Other Adverse Events (participants affected / at risk) | 0/381

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT04138576/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT04138576/ICF_001.pdf